CLINICAL TRIAL: NCT00764738
Title: Study Investigating High Resolution OCT, Multifocal ERG and Microperimetry Outcomes of Monthly vs As Needed Ranibizumab in Neovascular Age-Related Macular Degeneration
Brief Title: Study Investigating OCT, Multifocal ERG, and Microperimetry in Monthly Versus PRN Ranibizumab in Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Retina Macula Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4495s
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: ARMD; AMD; exudative AMD
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monthly (Active Comparator): Ranibizumab injections every month for 12 months.
  Interventions: Device: OCT, Multifocal ERG, Microperimetry; Drug: Ranibizumab Ophthalmic
- As Needed (Active Comparator): Ranibizumab injections monthly for 4 months then as needed thereafter.
  Interventions: Device: OCT, Multifocal ERG, Microperimetry; Drug: Ranibizumab Ophthalmic

INTERVENTIONS:
Device: OCT, Multifocal ERG, Microperimetry — OCT performed monthly. Fluorescein Angiography performed at baseline, month 3, month 5, month 8 and month 12.
  Microperimetry performed at baseline, month 3, month 5, month 8, and month 12 for monthly ranibizumab and at baseline, month 3, month 5 through month 12 for as needed ranibizumab.
  Multifocal ERG done at the same monthly visits as the microperimetry.
Drug: Ranibizumab Ophthalmic — 0.5 mg ranibizumab vs 2.0 mg ranibizumab

SUMMARY:
Visual outcomes using monthly ranibizumab therapy are well established in clinical trials, but the best way to assess when and how to treat patients with PRN therapy has not been proven. Information is lacking on Multi-focal ERG and microperimetry outcomes with ranibizumab therapy. Additionally, VA and OCT outcomes don't always correlate and other assessments such as the Multi-focal ERG and microperimetry may be useful as early predictors of when patients should be retreated. This study will assess 2 groups (monthly and PRN therapy) and assess high resolution OCT, microperimetry, and Multi-focal ERG outcomes. For the PRN group retreatment will be based on OCT criteria. We will investigate if microperimetry or multifocal ERG would have been an early predictor of fluid recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age greater or equal to 50 years old.
* Patients with active neovascular AMD

Exclusion Criteria:

* Pregnancy (Positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma)
* Previous PDT therapy
* Previous intravitreal steroid therapy within last 3 months
* Previous anti-VEGF therapy in the past month

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron P. Gallemore, MD, PhD, Principal Investigator — Retina Macula Institute
Locations (1):
- Retina Macula Institute, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Monthly Ranibizumab 0.5 mg: Intravitreal ranibizumab 0.5 mg dosing monthly for entire study.
- PRN Ranibizumab 0.5 mg: Intravitreal ranibizumab 0.5 mg dosing monthly for initial 4 injections followed by as needed dosing based on the presence of fluid on optical coherence tomography imaging.
- Monthly Ranibizumab 2.0 mg: Intravitreal ranibizumab 2.0 mg dosing monthly for entire study.
- PRN Ranibizumab 2.0 mg: Intravitreal ranibizumab 2.0 mg dosing monthly for initial 4 injections followed by as needed dosing based on the presence of fluid on optical coherence tomography imaging.
Period: Overall Study
Arm/Group | Monthly Ranibizumab 0.5 mg | PRN Ranibizumab 0.5 mg | Monthly Ranibizumab 2.0 mg | PRN Ranibizumab 2.0 mg
Started | 24 | 28 | 15 | 24
Completed | 22 | 25 | 12 | 18
Not Completed | 2 | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly Ranibizumab 0.5 mg | PRN Ranibizumab 0.5 mg | Monthly Ranibizumab 2.0 mg | PRN Ranibizumab 2.0 mg | Total
Number analyzed (Participants) | 22 | 25 | 12 | 18 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (1.0) | 75.8 (0.8) | 75.3 (1.4) | 78.8 (1.0) | 77.5 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 6 | 11 | 43
  Male | 11 | 10 | 6 | 7 | 34

OUTCOME MEASURES:

1. Primary Outcome: Multifocal Electroretinography N1-P1 Amplitude
Description: As measured within the central ring of the multifocal electroretinography study this measurement is the difference between the first positive peak (P1) and the first negative peak (N1).
Time Frame: One Year
Population: Required maintenance on device limited data collection for part of the study population.
Measure: Mean (Standard Error); unit: nV/deg^2
Groups:
- Monthly Ranibizumab: Intravitreal ranibizumab injections monthly for entire study.
- PRN Ranibizumab: Intravitreal ranibizumab injections monthly for initial 4 injections followed by as needed dosing based on the presence of fluid on optical coherence tomography imaging.
- Ranibizumab 0.5 mg: Intravitreal ranibizumab 0.5 mg dosing
- Ranibizumab 2.0 mg: Intravitreal ranibizumab 2.0 mg dosing.
Arm/Group | Monthly Ranibizumab | PRN Ranibizumab | Ranibizumab 0.5 mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 22 | 29 | 31 | 20
nV/deg^2
  Baseline | 3.6 (0.4) | 5.3 (0.4) | 4.9 (0.4) | 4.0 (0.4)
  1-year | 3.4 (0.4) | 4.7 (0.4) | 4.4 (0.4) | 3.6 (0.4)

2. Primary Outcome: Microperimetry Mean Sensitivity
Time Frame: One Year
Population: For 4 patients, data was unavailable on microperimetry from all visits (including screening).
Measure: Mean (Standard Error); unit: dB
Arm/Group | Monthly Ranibizumab | PRN Ranibizumab | Ranibizumab 0.5 mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 32 | 41 | 43 | 30
dB
  Baseline | 5.5 (0.8) | 5.1 (0.7) | 5.7 (0.7) | 4.6 (0.8)
  1-year | 6.7 (0.7) | 7.3 (0.8) | 7.3 (0.7) | 6.6 (1.0)

3. Secondary Outcome: Best Corrected Visual Acuity
Time Frame: One Year
Measure: Mean (Standard Error); unit: Letters
Arm/Group | Monthly Ranibizumab | PRN Ranibizumab | Ranibizumab 0.5 mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 34 | 43 | 47 | 30
Letters
  Baseline | 48.7 (4.0) | 52.6 (3.3) | 48.6 (3.5) | 54.5 (3.6)
  1-year | 56.4 (3.8) | 58.6 (3.4) | 55.4 (3.4) | 61.1 (3.6)

4. Secondary Outcome: Central Foveal Thickness on Optical Coherence Tomography
Time Frame: One Year
Measure: Mean (Standard Error); unit: micrometers
Arm/Group | Monthly Ranibizumab | PRN Ranibizumab | Ranibizumab 0.5 mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 34 | 43 | 47 | 30
micrometers
  Baseline | 341.2 (21.9) | 298.1 (16.8) | 308.2 (14.9) | 331.1 (26.2)
  1-year | 246.8 (17.0) | 227.9 (12.2) | 231.7 (14.3) | 242.7 (13.3)

ADVERSE EVENTS:
Arm/Group | Monthly Ranibizumab 0.5 mg | PRN Ranibizumab 0.5 mg | Monthly Ranibizumab 2.0 mg | PRN Ranibizumab 2.0 mg
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/25 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 1/22 | 2/25 | 0/12 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monthly Ranibizumab 0.5 mg (N=22) | PRN Ranibizumab 0.5 mg (N=25) | Monthly Ranibizumab 2.0 mg (N=12) | PRN Ranibizumab 2.0 mg (N=18)
Uveitic Glaucoma (Eye disorders) | NA | 1 | NA | NA
Vitreous Hemorrhage (Eye disorders) | NA | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monthly Ranibizumab 0.5 mg (N=22) | PRN Ranibizumab 0.5 mg (N=25) | Monthly Ranibizumab 2.0 mg (N=12) | PRN Ranibizumab 2.0 mg (N=18)
Corneal Abrasion (Eye disorders) | 0 | 1 | NA | NA
Injection Site Irritation (Eye disorders) | 1 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No